CLINICAL TRIAL: NCT04104230
Title: Quebec Pancreas Cancer Study
Acronym: QPCS
Status: Recruiting | Type: Observational
Sponsor: George Zogopoulos (Other)
Responsible Party: Sponsor-Investigator, George Zogopoulos, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 2018-3171
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Pancreas Neoplasm; Pancreas Cyst; Pancreatic Precancerous Condition; Familial Pancreatic Cancer; Hereditary Cancer; Bile Duct Cancer; Ampullary Cancer; Duodenal Cancer; Gallbladder Cancer
Keywords: Cancer Genetics
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst; Pancreatic carcinoma, familial; Bile Duct Neoplasms; Duodenal Neoplasms; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and/or saliva samples, tumor/tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Individuals Affected With Pancreatic Cancer: Individuals affected with pancreatic adenocarcinoma, with or without a family history of pancreatic adenocarcinoma.
- Individuals Affected with Related Cancer: Individuals affected with bile duct cancer, ampullary cancer, duodenal cancer or gallbladder cancer.
- Individuals Affected With Pancreatic Neoplasm: Individuals affected with pancreatic neoplasm, cyst or pre-cancerous lesion, with or without a family history of pancreatic adenocarcinoma.
- High-Risk Individuals: Individuals at high lifetime risk of pancreatic adenocarcinoma due to familial pancreatic cancer or hereditary cancer predisposition.
- Healthy Controls: Healthy individual at general population lifetime risk of pancreatic cancer and related cancers.

SUMMARY:
The Quebec Pancreas Cancer Study is a prospective clinic-based study consisting of clinical, family history and epidemiologic data, with accompanying biospecimens, from patients diagnosed with either pancreas cancer, a related cancer or a related pre-cancerous condition, and their families.

DETAILED DESCRIPTION:
The objectives of the QPCS are as follows:

1. To study the epidemiology of pancreas cancer, related cancers and related pre-cancerous conditions, including the risk factors and patient outcomes.
2. To characterize the contribution of known hereditary cancer syndromes to pancreas cancer, related cancers, and related pre-cancerous conditions.
3. To identify new genetic and epigenetic changes associated with hereditary pancreas cancer, related cancers, and related pre-cancerous conditions. DNA contains the instructions used in the development and functioning of living organisms, including humans. Epigenetic changes are changes other than changes in the underlying DNA sequence.
4. To study the tumour biology of pancreas cancer and related pre-cancerous conditions. This may include studying the tumour and the environment surrounding the tumour, as well as blood and/or saliva samples. The studies may include characterization of genetic, genomic, transcriptomic, epigenetic, proteomic, and metabolomic changes.
5. To identify and characterize biomarkers associated with pancreas cancer, related cancers and related pre-cancerous conditions.
6. To determine if there are any epidemiological, clinical and outcome (for example, overall survival) associations with the genetic, genomic, epigenetic, transcriptomic, proteomic, metabolomic or other biologic changes that occur in pancreas cancer, related cancers and related pre-cancerous conditions.

ELIGIBILITY:
Inclusion Criteria:

* Individual diagnosed with pancreatic cancer.
* Individual diagnosed with a related cancer (bile duct cancer, ampullary cancer, duodenal cancer, gallbladder cancer).
* Individual diagnosed with pancreatic neoplasm or pancreatic cyst.
* High-risk individuals with Familial Pancreatic Cancer (3 or more relatives affected with adenocarcinoma).
* High-risk individuals with 2 first-degree relatives affected with young-onset pancreatic adenocarcinoma (≤ 50 years old).
* High-risk individuals with one of the following Hereditary Cancer Syndromes: Peutz-Jeghers Syndrome (STK11 gene mutation), Familial Atypical Multiple Mole Melanoma Syndrome (CDKN2A gene mutation), or Hereditary Pancreatitis (PRSS1 gene mutation) with clinical manifestations.
* High-risk individuals with one of the following Hereditary Cancer Syndromes: Hereditary Breast and Ovarian Cancer Syndrome (BRCA1, BRCA2 or PALB2 gene mutation), Lynch Syndrome (MLH1, MSH2, MSH6, PMS2 or EPCAM gene mutation), or Hereditary Breast Cancer (ATM gene mutation), WITH a family history of cancer.

Exclusion Criteria:

* High-risk individuals with one of the following Hereditary Cancer Syndromes: Hereditary Breast and Ovarian Cancer Syndrome (BRCA1, BRCA2 or PALB2 gene mutation), Lynch Syndrome (MLH1, MSH2, MSH6, PMS2 or EPCAM gene mutation), or Hereditary Breast Cancer (ATM gene mutation), WITHOUT a family history of cancer.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with pancreatic cancer or related cancer followed in a hospital in Quebec.
  High-risk individuals with Familial Pancreatic Cancer or hereditary predisposition to pancreatic cancer with or without a family history of pancreatic cancer.
  Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-03-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge and Tissue Bank | 10 years
  Create a knowledge and tissue bank for pancreatic cancer, related pre-cancerous lesions, and related cancers, including patient demographics, type of chemotherapy treatments, type of surgical procedures, other procedures, overall survival, progression-free survival, epidemiological risk factors, genetic factors and characteristics of tumour tissue.

CONTACTS AND LOCATIONS:
Overall Officials: George Zogopoulos, MD, PhD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] Smith AL, Bascunana C, Hall A, Salman A, Andrei AZ, Volenik A, Rothenmund H, Ferland D, Lamoussenery D, Kamath AS, Amre R, Caglar D, Gao ZH, Haegert DG, Kanber Y, Michel RP, Omeroglu-Altinel G, Asselah J, Bouganim N, Kavan P, Arena G, Barkun J, Chaudhury P, Gallinger S, Foulkes WD, Omeroglu A, Metrakos P, Zogopoulos G. Establishing a clinic-based pancreatic cancer and periampullary tumour research registry in Quebec. Curr Oncol. 2015 Apr;22(2):113-21. doi: 10.3747/co.22.2300. PMID 25908910
- [Background] Andrei AZ, Hall A, Smith AL, Bascunana C, Malina A, Connor A, Altinel-Omeroglu G, Huang S, Pelletier J, Huntsman D, Gallinger S, Omeroglu A, Metrakos P, Zogopoulos G. Increased in vitro and in vivo sensitivity of BRCA2-associated pancreatic cancer to the poly(ADP-ribose) polymerase-1/2 inhibitor BMN 673. Cancer Lett. 2015 Aug 1;364(1):8-16. doi: 10.1016/j.canlet.2015.04.003. Epub 2015 Apr 9. PMID 25864590
- [Background] Smith AL, Alirezaie N, Connor A, Chan-Seng-Yue M, Grant R, Selander I, Bascunana C, Borgida A, Hall A, Whelan T, Holter S, McPherson T, Cleary S, Petersen GM, Omeroglu A, Saloustros E, McPherson J, Stein LD, Foulkes WD, Majewski J, Gallinger S, Zogopoulos G. Candidate DNA repair susceptibility genes identified by exome sequencing in high-risk pancreatic cancer. Cancer Lett. 2016 Jan 28;370(2):302-12. doi: 10.1016/j.canlet.2015.10.030. Epub 2015 Nov 3. PMID 26546047
- [Background] Smith AL, Wong C, Cuggia A, Borgida A, Holter S, Hall A, Connor AA, Bascunana C, Asselah J, Bouganim N, Poulin V, Jolivet J, Vafiadis P, Le P, Martel G, Lemay F, Beaudoin A, Rafatzand K, Chaudhury P, Barkun J, Metrakos P, Marcus V, Omeroglu A, Chong G, Akbari MR, Foulkes WD, Gallinger S, Zogopoulos G. Reflex Testing for Germline BRCA1, BRCA2, PALB2, and ATM Mutations in Pancreatic Cancer: Mutation Prevalence and Clinical Outcomes From Two Canadian Research Registries. JCO Precis Oncol. 2018 Nov;2:1-16. doi: 10.1200/PO.17.00098. PMID 35135108
- [Background] Li Q, Wang H, Zogopoulos G, Shao Q, Dong K, Lv F, Nwilati K, Gui XY, Cuggia A, Liu JL, Gao ZH. Reg proteins promote acinar-to-ductal metaplasia and act as novel diagnostic and prognostic markers in pancreatic ductal adenocarcinoma. Oncotarget. 2016 Nov 22;7(47):77838-77853. doi: 10.18632/oncotarget.12834. PMID 27788482
- See also: QPCS Website — http://www.cancerpancreas.ca/